CLINICAL TRIAL: NCT03504592
Title: Utilizing mHealth to Improve Diabetes in an Obstetric Population
Brief Title: Smartphone Utilization for Glucose Monitoring and Antenatal Reporting
Acronym: SUGAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Lisa Gray, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00068149
Record Dates: First submitted 2018-03-09; First posted 2018-04-20 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Gestational Diabetes; Pregestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glooko App (Experimental): Glooko application and meter compatibility device (if required)
  Interventions: Behavioral: Completion of Glucose logs
- Traditional Care (Active Comparator): Traditional clinic reporting system: paper/MyChart/emailed glucose logs
  Interventions: Behavioral: Completion of Glucose logs

INTERVENTIONS:
Behavioral: Completion of Glucose logs — Glucose logs will be assessed by provider for completeness and accuracy

SUMMARY:
This project will utilize MHealth technology to address the barriers providers and obstetric patients experience when reporting blood glucose results. Half of the participants will record their blood glucose values with the assistance of a smartphone device, the other half will continue in the traditional care method of the clinic.

DETAILED DESCRIPTION:
This will be a prospective single center randomized trial piloting the use of mHealth applications in an obstetric population with diabetes. Participants will be enrolled in the study after the diagnosis of diabetes is made in pregnancy for those with gestational diabetes, or for patients with preexisting diabetes they will be enrolled upon initiation of prenatal care. Participants will be randomized to traditional care or mHealth intervention. Outcomes will include completeness and accuracy of the participant glucose log, unscheduled health care access episodes in the pregnancy, patient satisfaction, percentage of glucose values at goal and percent change in Hemoglobin A1C.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, English speaking, Diagnosed with diabetes during pregnancy or with known preexisting diabetes, has smartphone, sees URMC OBGYN for obstetric care in pregnancy.

Exclusion Criteria:

* Not English speaking, does not have smartphone, unable to consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients must be pregnant to be enrolled in this study
Enrollment: 21 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Completeness and accuracy of blood glucose record | Every 2 weeks through study completion, up to 42 weeks
  The number of values reported to the provider out of the number that should have been collected during the time period, expressed as a percent, as well as the number of values reported that were verified accurate by the meter out of the total number of values reported in the time frame expressed as a percent.

SECONDARY OUTCOMES:
Patient Satisfaction | Once prior to exiting the study, an average of 42 weeks
  Responses to patient satisfaction survey
Glucose values at goal | Every 2 weeks through study completion, up to 42 weeks
  % of glucose values at goal during the study period
% Change in Hemoglobin A1C | Once prior to exiting the study, up to 42 weeks
  % of change in values of HbA1C during the study period
Clinic visits | through study completion, up to 42 weeks
  Number of clinic visits during the study period
Unscheduled health care access episodes | through study completion, up to 42 weeks
  Number of unanticipated or unscheduled health care visits during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- UR Medicine Obstetrics and Gynecology, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided